CLINICAL TRIAL: NCT02844777
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Cohort Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Once-Daily Application of Topical VDA-1102 Ointment for 28 Days in Subjects With Actinic Keratosis
Brief Title: Efficacy and Safety of VDA-1102 Ointment in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vidac Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VDA-CP-03
Record Dates: First submitted 2016-06-29; First posted 2016-07-26 (Estimated); Results first posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2021-05

CONDITIONS: Actinic Keratosis
Keywords: topical ointment; skin; hexokinase; precancerous conditions; carcinoma, squamous cell
MeSH Terms: conditions — Keratosis, Actinic; Precancerous Conditions; Carcinoma, Squamous Cell | interventions — Excipients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Excipeint alone
  Interventions: Drug: Placebo
- 5% VDA-1102 (Experimental): Active study medication
  Interventions: Drug: 5% VDA-1102
- 10% VDA-1102 (Experimental): Active study medication
  Interventions: Drug: 10% VDA-1102

INTERVENTIONS:
Drug: Placebo — 200 mg applied once-daily for 28 days
  Other Names: Excipients alone; Matched-placebo
  Arms: Placebo
Drug: 5% VDA-1102 — 200 mg applied once-daily for 28 days
  Other Names: 5% VDA-1102 topical dermal ointment
  Arms: 5% VDA-1102
Drug: 10% VDA-1102 — 200 mg applied once-daily for 28 days
  Other Names: 10% VDA-1102 topical dermal ointment
  Arms: 10% VDA-1102

SUMMARY:
This Phase 2 clinical trial is a multi-center, randomized, double-blind, placebo-controlled, multiple-dose, parallel-cohort study to assess the efficacy, safety and tolerability of VDA-1102 in the treatment of actinic keratosis (AK) on the head of male and female adult subjects.

DETAILED DESCRIPTION:
Approximately 84 subjects who meet the study's enrollment criteria at the completion of the Screening Period will be randomized to receive 5% or 10% VDA-1102, or matched-placebo. During the Treatment Period, study drug will be applied once-daily for 28 days to a 25 square centimeter area of skin containing 4-8 actinic keratosis lesions on the face or scalp. Subjects will be followed for an additional 28 days (Observation Period) wherein no study drug will be applied.

The purpose of the study is to determine whether once-daily application of VDA-1102 ointment for 28 days is effective and well-tolerated in the treatment of actinic keratosis of the face and scalp.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject has a minimum of 4 and a maximum of 8 discrete Grade 1-2 AK lesions within a single 25 square centimeter area of skin on their scalp or face

Main Exclusion Criteria:

* Subject is: (a) pregnant; (b) lactating; (c) planning to become pregnant during the study, or (d) fertile and they or their fertile partner is unable or unwilling to use the required contraceptive methods
* Subject is immunosuppressed
* Subject has used any of the following topical treatments in the Treatment Field: (1) topical retinoids within 8 weeks of Screening or (2) micro-dermabrasion, laser ablative treatments, ALA-PDT, chemical peels, 5-FU, diclofenac, imiquimod, ingenol, or other topical treatments for AK or that might impact AK within 12 weeks of Screening.
* Subject has used systemic retinoid therapy within 6 months of Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaim M Brickman, MD, Study Director — Vidac Pharma
Locations (1):
- Therapeutics Clinical Research, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 5% VDA-1102 | 10% VDA-1102
Started | 29 | 32 | 32
Completed | 27 | 32 | 32
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 5% VDA-1102 | 10% VDA-1102 | Total
Number analyzed (Participants) | 29 | 32 | 32 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (7.8) | 67.3 (8.2) | 66.3 (11.8) | 66.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 29 | 83
  Male | 3 | 4 | 3 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 27 | 80
  Israel | 3 | 5 | 5 | 13
Fitzpatrick skin types [Count of Participants; unit: Participants]
  I : Pale white skin, always burns, and never tans | 5 | 4 | 6 | 15
  II : White skin, usually burns easily, tans minimall | 17 | 18 | 24 | 59
  III : Light brown skin, burns moderately, tans uniformly | 7 | 9 | 2 | 18
  IV : Moderate brown skin, burns minimally, always tans well. | 0 | 1 | 0 | 1
Treatment field location [Count of Participants; unit: Participants]
  Face | 23 | 24 | 23 | 70
  Scalp | 6 | 8 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Actinic Keratosis Lesions in the Treatment Field on Day 56
Description: To compare the reduction on Day 56 in the number of the actinic keratosis (AK) lesions in the Treatment Field of subjects receiving once-daily topical 5% or 10% VDA-1102 ointment for 28 days to the reduction in the number of AK lesions in subjects receiving placebo.
Time Frame: Baseline and day 56
Population: ITT
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo | 5% VDA-1102 | 10% VDA-1102
Number analyzed (Participants) | 26 | 32 | 32
lesions | -1.54 (1.79) | -1.34 (1.98) | -1.94 (1.97)
Statistical Analysis 1: Comparison: Placebo vs 5% VDA-1102; Test type: Other; p = 0.9518, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 10% VDA-1102; Test type: Other; p = 0.2458, ANCOVA

2. Other Pre Specified Outcome: Percentage of Patients With Complete Clearance of Actinic Keratosis Lesions in the Treatment Field
Description: The percentage of subjects achieving complete clearance of AK lesions within the Treatment Field on Day 56.
Time Frame: Baseline and Day 56
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 5% VDA-1102 | 10% VDA-1102
Number analyzed (Participants) | 26 | 32 | 32
Participants | 1 | 3 | 2
Statistical Analysis 1: Comparison: Placebo vs 5% VDA-1102; Test type: Other; p = 0.6201, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs 10% VDA-1102; Test type: Other; p = 1.0000, Fisher Exact

3. Other Pre Specified Outcome: Change From Baseline in the Number of AK Lesions Within the Treatment Field of Each Subject on Day 84.
Description: To compare the reduction on Day 84 in the number of the actinic keratosis lesions
Time Frame: Baseline and day 84
Population: ITT population
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo | 5% VDA-1102 | 10% VDA-1102
Number analyzed (Participants) | 14 | 20 | 20
lesions | -1.64 (1.69) | -2.05 (1.82) | -2.15 (2.01)
Statistical Analysis 1: Comparison: Placebo vs 5% VDA-1102; Test type: Other; p = 0.2912, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 10% VDA-1102; Test type: Other; p = 0.4168, ANCOVA

4. Other Pre Specified Outcome: AK Grade 2 Lesions Number: Change From Baseline (Day 1 Pre-dose) in Sub-group of Subjects With at Least One Grade 2 Lesion at Baseline (From ITT Population)
Description: Change from Baseline (Day 1 Pre-dose) in Sub-group of Subjects with at least one Grade 2 Lesion at Baseline (from ITT Population)in the number of grade ≥ 2 lesions.
  Grade 2 defined as: moderate (moderately thick AK that are easily seen and felt)
Time Frame: Baseline and day 56
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo | 5% VDA-1102 | 10% VDA-1102
Number analyzed (Participants) | 20 | 27 | 22
lesions | -1.20 (1.99) | -1.00 (2.08) | -2.50 (2.44)
Statistical Analysis 1: Comparison: Placebo vs 5% VDA-1102; Test type: Other; p = 0.6458, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 10% VDA-1102; Test type: Other; p = 0.0721, ANCOVA

5. Other Pre Specified Outcome: Change From Baseline in the Adjusted Number of Lesions Weighted by Grade ([Number of Grade 1 Lesions] + [2× Number of Grade 2 Lesions] + [3× Number of Grade 3 Lesions])
Description: Change From Baseline in the Adjusted Number of Lesions Weighted by Grade ([Number of Grade 1 Lesions] + [2× Number of Grade 2 Lesions] + [3× Number of Grade 3 Lesions]) Grade 1 - mild (slightly palpable AK that are felt better than seen) Grade 2 - moderate (moderately thick AK that are easily seen and felt) Grade 3 - severe (very thick and/or obvious AK).
Time Frame: Baseline and day 56
Population: ITT population
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo | 5% VDA-1102 | 10% VDA-1102
Number analyzed (Participants) | 26 | 32 | 32
lesions | -27.8 (35.6) | -24.6 (40.5) | -38.5 (35.3)
Statistical Analysis 1: Comparison: Placebo vs 5% VDA-1102; Test type: Other; p = 0.4200, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 10% VDA-1102; Test type: Other; p = 0.0241, ANCOVA

ADVERSE EVENTS:
Time Frame: Screening to Day 84
Arm/Group | Placebo | 5% VDA-1102 | 10% VDA-1102
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/32 | 1/32
Other Adverse Events (participants affected / at risk) | 3/29 | 1/32 | 4/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=29) | 5% VDA-1102 (N=32) | 10% VDA-1102 (N=32)
benign sero-mucinous cystadenoma of abdomen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=29) | 5% VDA-1102 (N=32) | 10% VDA-1102 (N=32)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/77/NCT02844777/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT02844777/SAP_001.pdf